CLINICAL TRIAL: NCT04640727
Title: ORIF Versus CRIF of Completely Displaced and Rotated Lateral Condylar Fractures of the Humerus in Children：a Ambispective Chort Study
Brief Title: ORIF Versus CRIF of Completely Displaced and Rotated Lateral Condylar Fractures of the Humerus in Children
Status: Enrolling by invitation | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Hongwen Xu, Guangzhou Women and Children's Medical Center, Guangzhou Women and Children's Medical Center
Other Study IDs: GuangzhouWCMC-004
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Humeral Fractures
Keywords: Open reduction and internal fixation; Closed reduction and internal fixation; completely displaced and rotated lateral condylar fracture
MeSH Terms: conditions — Humeral Fractures | interventions — Open Fracture Reduction; Closed Fracture Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- open reduction and internal fixation: open reduction and internal fixation used in treating completely displaced and rotated lateral condylar fracture in children
  Interventions: Procedure: open reduction
- closed reduction and internal fixation: closed reduction and internal fixation used in treating completely displaced and rotated lateral condylar fracture in children
  Interventions: Procedure: closed reduction

INTERVENTIONS:
Procedure: open reduction — A sterile tourniquet is applied and an oblique posterolateral skin incision is made. Superficial dissection is carried out in the plane of the fracture hematoma until the distal lateral corner of the proximal fragment is identified. Once the metaphyseal side of the fracture has been identified, the dissection is carried across the joint to expose the medial articular surface. After exposure of the proximal fragment, the orientation of the distal fragment is defined and the soft tissues are sharply released off the anterior aspect of the distal fragment, with extension carried distally to the radial head. After irrigation and débridement of the fracture hematoma, the distal fragment is reduced with a towel clip. It is important to judge the reduction at the level of the articular surface rather than the metaphysis because plastic deformation or comminution of the metaphyseal fragment may be present. Pins (usually 0.062 inch) are placed percutaneously to secure the fracture.
  Groups: open reduction and internal fixation
Procedure: closed reduction — we applied a gentle varus force to the elbow while the patient was under general anesthesia, and we attempted to reposition the rotated fragment by directly pushing or by using Kirschner wires as joysticks . After repositioning, we applied gradual direct compression to the distal fracture fragment anteromedially.We then applied slight valgus force to the elbow with the forearm supinated and the elbow fully extended to maintain the reduction. After the fracture reduction was confifirmed to be within 2 mm, especially as seen on the anteroposterior, lateral radiographs,and internal obliquewe used smooth Kirschner wires to perform percutaneous pinning
  Groups: closed reduction and internal fixation

SUMMARY:
Open reduction and internal fixation has been widely used in treating completely displaced and rotated lateral condylar fracture in children and it usually produces good results. Only a few studies reported Closed reduction and internal fixation is an effective treatment for completely displaced and rotated lateral condyle fractures of the humerus, but evidence on its effectiveness and safety is scarce. The aim of the trial was to compare functional and outcome use in patients treated completely displaced and rotated lateral condylar fracture with ORIF versus CRIF.

DETAILED DESCRIPTION:
Lateral condylar humerus fractures are the second most common elbow fracture in children, accounting for approximately 17-20% of pediatric elbow fractures. Jakob et al. first described a novel classification based on the presence of cartilage bridging. It was modified by Foster et al. who identified the differences in outcomes between fractures with < 2 mm and ≥ 2 mm displacement. most surgeons preferred open reduction and internal fixation (ORIF) to insure anatomic reduction of these unstable intra-articular fractures. Only a few reports have focused on closed reduction and Percutaneous Pinning (CRPP) of lateral condylar humeral fractures. In most studies, this technique was used only in cases with displacement between 2 and 4mm. CRPP has shown several advantages over ORIF, including less dissection of soft tissue around the fragment, low risk of vessel damage, low risk of non-union and avascular necrosis (AVN) of distal humerus physeal, shorter operating room times, and avoidance of an open incision with an unaesthetic scar. Song et al. introduced a new classification and an internal oblique view to better assess the displacement of the fragment, and they managed to achieve closed reduction of the fracture, even in cases with displacement exceeding 4mm or those with rotational displacement (graded as stage 5 according Song classification and Type III according to Jakob classification). Because the study was not controlled, we could not tell the difference between cases treated with CRPP and the cases treated with ORIF directly.

Since May 1, 2019, at our Institution, we have been treating type III lateral condyle fractures with CRPP. The primary objective of this study was to report the efficacy and safety of CRPP of lateral condyle fracture. The secondary aim was to compare the outcomes between CRPP and ORIF.

ELIGIBILITY:
Inclusion Criteria:

* completely displaced and rotated lateral condyle fractures of the humerus (Jakob Stage 3)

Exclusion Criteria:

- presented more than 7 days after the fracture , Capitulum humerus cannot be clearly identified on X-ray， had experienced a previous lateral condyle fractures on the same limbs, pathological fracture， open fracture， Combined with other fractures at the same time，

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: After Internal Review Board approval, all Type III lateral condyle fractures according to Jakob classification were reviewed at our institution from 2017 to 2021
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Hardacre criteria | 1 years follow up
  Excellent：No limitation of Range of Motion， No alteration of Carrying Angle，No symptoms Good： Functional range of motion (lacking no more 15" of complete extension)，Inconspicuous alteration of Carrying Angle，No arthritic and neurologic symptoms Poor：Disabling loss of function， Conspicuous alteration of Carrying Angle，have Arthritic symptom, ulnar neuritis, roentgen findings of nonunion, avascular necrosis

SECONDARY OUTCOMES:
duration of operation | during the operation
  From TIME OUT to long-arm cast immobilization completed
amount of bleeding | during the operation
  From TIME OUT to long-arm cast immobilization completed
Radiation exposure | during the operation
  From TIME OUT to long-arm cast immobilization completed
The interepicondylar width (IEW) | 3 months after the surgery
  The interepicondylar width (IEW) has previously been described to quantify the magnitude of lateral spurring. The IEW was measured on the initial injury radiograph as well as the postoperative radiograph obtained approximately 3 months after surgery. The magnitude of lateral spurring, expressed as a ratio of the postoperative to the injury IEW, was defined as normal if it was <1.05, mild spurring from 1.05 to 1.1, moderate spurring from 1.1 to 1.2, and severe spurring >1.2

CONTACTS AND LOCATIONS:
Overall Officials: Hongwen Xu, doctor, Principal Investigator — Guangzhou Women & Children Medical Center
Locations (1):
- Guangzhou Women & Children Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No